CLINICAL TRIAL: NCT02442804
Title: The Effects of Pomegranate Polyphenols on Neuropsychological Functioning Following Ischemic Stroke
Brief Title: Cognitive Impact of Pomegranate Polyphenols Following Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, John Bellone, MA, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5150112
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: Pomegranate; Stroke; Neuropsychology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke - POMx (Experimental): Pomegranate supplement (1g) by mouth twice per day for 7 days
  Interventions: Dietary Supplement: POMx
- Stroke - Placebo (Placebo Comparator): Placebo (for POMx, containing no antioxidant contents; 1g) capsule by mouth twice per day for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: POMx — Pomegranate supplement (1g) by mouth twice per day for 7 days
  Arms: Stroke - POMx
Other: Placebo — Placebo (for POMx, containing no antioxidant contents; 1g) capsule by mouth twice per day for 7 days
  Arms: Stroke - Placebo

SUMMARY:
The purpose of this study is to determine whether pomegranate supplements improve cognitive functioning following stroke.

DETAILED DESCRIPTION:
Research suggests that antioxidants (substances that may slow or prevent cell damage) found in many fruits and vegetables may help improve brain functioning (for example, memory and attention) in healthy individuals and prevent cognitive decline in individuals who have suffered a stroke. The purpose of this research study is to examine whether dietary supplementation with an antioxidant extract can help promote healthy cognitive functioning as a component of recovery after stroke. The procedures include: Administering polyphenols via 2 POMx pills, each of which contains polyphenols derived from pomegranates equivalent to the content of approximately 8 ounces of pomegranate juice, or placebo pills (capsules containing no polyphenol ingredients), every day for one week to inpatients who are in the acute post-stroke phase. Neuropsychological testing pre- and post-treatment will determine whether cognitive functioning changes. Subjects will be randomized into either a placebo or polyphenol group.

ELIGIBILITY:
Inclusion Criteria:

* Suffered an ischemic stroke and admitted to LLUMC Rehabilitation Institute for inpatient care
* Fluent in English
* Between the age of 18 and 89 years old

Exclusion Criteria:

* Less than 6 years of education
* Global aphasia
* Pregnant
* History of allergy to pomegranates
* History of traumatic brain injury
* Neurodegenerative disease or neurologic condition with known cognitive impact (e.g., Alzheimer's disease)
* Active renal disease
* Active liver disease
* Intracerebral hemorrhage in past 6 months
* Neurosurgery in past month
* Taking warfarin (Coumadin)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University East Campus Hospital, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stroke - POMx | Stroke - Placebo
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke - POMx | Stroke - Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.13 (13.62) | 59.63 (13.48) | 58.88 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 4 | 5 | 9
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Score
Description: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) provides both a total scale score and scores for 5 different cognitive domains. It is relatively brief (approximately 20 minutes total) and has alternate forms. Specifically, the test measures immediate memory (with list learning and story memory), visuospatial/constructional ability (with figure copy and line orientation), language (with picture naming and semantic fluency), attention (with digit span and coding), and delayed memory (with list recall, list recognition, story recall, and figure recall). Scores from all subtests are aggregated into a total composite score (manual provides conversion procedure). RBANS data were age-normed based on the sample described in the manual (Randolph, 2012) and were analyzed as index scores (also referred to as standard scores), which have a mean of 100 and a standard deviation of 15. Higher scores on each sub measure and index indicate better performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: standard score change
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
standard score change | 6.86 (6.52) | 1.29 (6.65)

2. Secondary Outcome: Change From Baseline Mini-Mental State Examination - 2nd Edition Score
Description: The MMSE-2 is a brief (about 10 minutes) screening tool that touches upon orientation to time and place, recall, attention/calculation, naming, repetition, comprehension, reading, writing, and drawing, with all the scores from these domains cumulating to a maximum of 30 points (minimum = 0). Higher score indicates better performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
raw score | 0.83 (2.48) | 0.43 (2.64)

3. Secondary Outcome: Change From Baseline Functional Independence Measure (FIM) Score
Description: Functional Independence Measure (FIM) Score consists of eighteen sub-measures under the following 6 categories: Self-Care (eating, grooming, bathing, dressing upper body, dressing lower body, toileting), Sphincter Control (bladder control, bowel control), Transfers (bed/chair/wheelchair transfer, toilet transfer, tub/shower transfer), Locomotion (walk/wheelchair, stairs), Communication (comprehension, expression), and Social Cognition (social interaction, memory, problem solving). Scores for each sub-measure range from 1 (total assistance) to 7 (complete independence), and the 18 scores are summed to obtain the FIM score. Higher scores indicate better performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 8 | 8
raw score | 22.63 (15.17) | 7.25 (6.82)

4. Secondary Outcome: Change From Baseline Trail-making Test Part A Score
Description: The Trail-making Test consists of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. Results for the test are reported as the number of seconds required to complete the task (ranges from 0 to 300; discontinued at 300 seconds); therefore, higher scores reveal greater impairment.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
seconds | -18.14 (18.8) | -19.86 (33.35)

5. Secondary Outcome: Change From Baseline Brief Test of Attention Score
Description: On the Brief Test of Attention (BTA), the examinee listens to a string of numbers and letters and must mentally tally (without the use of their fingers) how many numbers are in a particular trial. They do this for 10 trials and then are given 10 additional trials with the task of tallying how many letters they hear. The task increases in difficulty as the trials progress, and the entire test takes 5-10 minutes to complete. The scorer adds the number of trials correct from all 20 trials to attain a total score (ranges from 0 to 20). Higher scores indicate better performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
raw score | 3.29 (1.38) | 0.14 (2.41)

6. Secondary Outcome: Change From Baseline Controlled Oral Word Association Test Score
Description: The Controlled Oral Word Association Test (COWAT) is a measure of controlled verbal fluency that involves the examinee naming as many words that begin with a certain letter of the alphabet as he or she can in 1 minute. There are a few rules (i.e., no proper nouns and no words that have the same meaning and only differ by its suffix) and the task is repeated twice more with different letters each time. The scorer tallies the total acceptable words from all 3 trials into one total score (ranges from 0 on up). Higher total score indicates better performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: number of acceptable words
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
number of acceptable words | 1.29 (2.43) | 2.14 (3.67)

7. Secondary Outcome: Change From Baseline Line Bisection Test Score
Description: The Line Bisection Test consists of 20 horizontal lines of varying length and proximity to the center of a sheet of paper (i.e., some are closer to the left or right sides of the page). The examinee is asked to place a mark to bisect each line. The scorer measures the degree of deviation from the center of each line (in cm) and attains the absolute value of the average percentage of deviation across all 20 lines. The scorer also attains the dominant direction of deviation (i.e., whether the examinee misses more to the left or to the right on average across the 20 lines). The value of the largest deviation is imputed for any omissions. Percentage ranges from 0 on up. Higher percentage of deviation indicates worse performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: percentage of deviation from center
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
percentage of deviation from center | -0.91 (3.79) | -3.71 (4.69)

8. Secondary Outcome: Change From Baseline Trail-making Test Part B Score
Description: The Trail-making Test Part B consists of circles with either numbers (1 - 13) or letters (A - L) in them; as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). Results for both TMT A and B are reported as the number of seconds required to complete the task (ranges from 0 to 300; discontinued at 300 seconds); therefore, higher scores reveal greater impairment.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
seconds | -20 (21.03) | -39 (39.64)

9. Secondary Outcome: Change From Baseline Animals Fluency Score
Description: The Animal Fluency task involves providing the examinee a category prompt. For example, the examiner asks the examinee to name as many animals as he or she can in 1 minute. The total number of acceptable words is tallied for a total score (ranging from 0 on up). Higher scores indicate better performance.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: number of acceptable words (animals)
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
number of acceptable words (animals) | -0.14 (2.19) | 3.14 (2.67)

10. Secondary Outcome: Change From Baseline Beck Depression Inventory - II (BDI-II) Score
Description: The Beck Depression Inventory - Second Edition (BDI-II) is a widely used self-report questionnaire of depressive symptoms. The examinee is asked to respond to 21 items by endorsing whether or not they experience symptoms of sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping pattern, irritability, changes in appetite, concentrating difficulty, tiredness or fatigue, and loss of interest in sex. Examinees can also describe the degree of severity of each symptom, as each item ranges from 0-3. The scorer adds the scores for each item to attain a total score, which is interpreted according to the following guidelines: 0-13 = minimal depression, 14-19 = mild depression, 20-28 = moderate depression, 29-63 = severe depression
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
raw score | 0.14 (9.58) | -3.86 (9.48)

11. Secondary Outcome: Change From Baseline State-Trait Anxiety Inventory - State Score
Description: The State-Trait Anxiety Inventory (STAI) is a self-report inventory of anxiety symptoms. The test consists of two parts: 20 questions that assess anxiety level at the time of the examination (i.e., state) and 20 questions that assess the examinee's general level of anxiety (i.e., trait). Items include feeling at ease, feeling upset, feeling self-confident, feeling confused, feeling like a failure, feeling rested, and having disturbing thoughts, among others. Examinees endorse 1 of 4 options on a likert scale, from "not at all" to "very much so." Each of the scales (state and trait) ranges from 0 to 80. Higher score indicates more anxiety symptoms.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
raw score | -5.86 (10.43) | -2.86 (12.62)

12. Secondary Outcome: Change From Baseline State-Trait Anxiety Inventory - Trait Score
Description: as for outcome 11
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Stroke - POMx | Stroke - Placebo
Number analyzed (Participants) | 7 | 7
raw score | -1.57 (7.87) | -1 (9.17)

ADVERSE EVENTS:
Arm/Group | Stroke - POMx | Stroke - Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stroke - POMx (N=8) | Stroke - Placebo (N=8)
Psychotic Episode (Psychiatric disorders) | 1 (1) | 0 (0) — The participant experienced auditory hallucinations and a psychiatry consultant recommended withdrawal from the experiment. Notably, this subject began experiencing auditory hallucinations several days prior to POM administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No